CLINICAL TRIAL: NCT06921356
Title: Groceries Plus Multi-Component Lifestyle Intervention for Adults With Hypertension and Type 2 Diabetes Residing in Urban Food Deserts (DASH-Life): Pilot Randomized Clinical Trial
Brief Title: Groceries Plus Multi-Component Lifestyle Intervention for Adults With Hypertension and Type 2 Diabetes
Acronym: DASH-Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00425074; P50MD017348 (NIH)
Record Dates: First submitted 2025-03-31; First posted 2025-04-10 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus (T2DM)
Keywords: hypertension; type 2 diabetes; diet
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Shopping DASH diet advice group (S-DASH) (Active Comparator)
  Interventions: Behavioral: Self-Shopping DASH diet advice
- Coach-Directed Tailored DASH Groceries Plus Lifestyle Intervention (C-DASH) (Experimental)
  Interventions: Behavioral: Coach-Directed Tailored DASH Groceries Plus Lifestyle Intervention

INTERVENTIONS:
Behavioral: Coach-Directed Tailored DASH Groceries Plus Lifestyle Intervention — Participants assigned to the C-DASH group will meet by telephone with the study coach for 1 hour, and then have brief weekly conversations (about 15-30 minutes) by phone during the first three months. During these weekly calls, the study coach will assist participant with selecting fruits, vegetables, nuts, and beans. During months 4-6, the study coach will continue to work with participant to set goals for following the DASH-Life way of eating, but the study will no longer provide a weekly food allowance to purchase groceries.
  Arms: Coach-Directed Tailored DASH Groceries Plus Lifestyle Intervention (C-DASH)
Behavioral: Self-Shopping DASH diet advice — Participants assigned to the S-DASH group will receive a brochure about the DASH eating plan. For the first three months, Participants will also receive a gift card to shop at a local supermarket. During months 4-6, participants will be asked to continue following the DASH eating plan listed in the brochure but will no longer be provided the grocery gift card.
  Arms: Self-Shopping DASH diet advice group (S-DASH)

SUMMARY:
People with high blood pressure and diabetes often have low levels of key nutrients as a result of not eating enough fresh fruits and vegetables. Research studies suggest that these nutrients can lower blood pressure and blood sugar. This study will investigate if providing encouragement to adopt this healthy and nutritious way of eating and providing guidance on weight management will lower blood pressure and blood sugar. The DASH-Life research study will recruit adults with hypertension and type 2 diabetes who live in Baltimore metro areas that don't have many stores selling healthy foods. The DASH-Life research study is 6 months long. Participants will be randomly assigned to one of two groups: 1) Self-Shopping DASH (S-DASH) diet advice group, or 2) Coaching DASH (C-DASH) diet advice group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diabetes Mellitus Type 2 defined by: self-reported type 2 diabetes diagnosis, or HbA1c>=6.5%, or treatment of diabetes with diabetes medications(s)
* Baseline systolic BP 120-159 mmHg (with or without medications.)
* Serum potassium level >3.0 and <5 mmol/L,
* Estimated glomerular filtration rate (eGFR) >=45 mL/min/1.73m2.
* Willing and able to complete required procedures in English.
* Living in Healthy Food Priority Area in Baltimore; the US Department of Agriculture (USDA) defined low income, low access areas, or census blocks with area deprivation index (ADI) 60 and above (State Decile>=6.)

Exclusion Criteria:

* Hypoglycemia requiring hospitalization or the assistance of another person in the last 6 months
* Cardiovascular event within 6 months
* On diabetes or weight loss medications such as glucagon-like peptide 1 (GLP-1), GLP-1/glucose-dependent insulin-releasing peptide (GIP), insulin, or any combination of these medications
* HbA1c ≥ 10%
* Type 1 diabetes
* Baseline systolic BP < 100 mmHg
* Weight >400 lbs due to the maximum weight on study scale
* Chronic disease that might interfere with trial participation
* Current participation in another clinical trial that might affect blood pressure, weight loss, diabetes, or ability to adhere to study procedures
* Current participation in program with conflicting dietary guidance (i.e., meal replacement or keto diets)
* Unwillingness or inability to adopt a DASH-like diet
* Planning to leave area in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by the number of participants enrolled | Baseline
  The observed count of responses to the prescreening will be summarized. Recruitment yields at screening visit and randomization visit will be derived.
Acceptability as assessed by the Acceptability of the Intervention Measure survey | 3 months
  Acceptability of the intervention will be quantitatively measured by the Acceptability of Intervention Measure (AIM) survey. The survey consists of 4 items, each measured on a 5-point Likert scale from 1 (completely disagree) to 5 (completely agree). The score is calculated as the mean of the responses to the 4 items. A higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yeh, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth Clinical Research Unit, Baltimore, Maryland, United States